CLINICAL TRIAL: NCT05892029
Title: Using Machine Learning Algorithms to Develop a Risk Prediction Model for Phthalate-ester-induced Diseases and Suggestions for Improved Nursing Assessment
Brief Title: Develop a Risk Prediction Model for Phthalate-ester-induced Diseases
Status: Completed | Type: Observational
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Pei-Hung Liao, Associate Professor, National Taipei University of Nursing and Health Sciences
Other Study IDs: (862)110-08
Record Dates: First submitted 2023-05-19; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Plasticizers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This exploratory study collected basic demographic and laboratory data from the Taiwan Biobank using artificial intelligence algorithms and applied data mining to identify the correlations between phthalate esters [di(2-ethylhexyl) phthalate, DEHP], lifestyle, and disease.

DETAILED DESCRIPTION:
This study was designed as exploratory research. The Institutional Review Board and the Taiwan Biobank approved the study before it was conducted (Approval Number: TWBR11007-06). The data set included information from participants between 30 and 70 years old who were tested for PAEs between 2016 and 2022 (1337 cases). The data set includes (1) questionnaire responses, such as basic personal information, individual health behaviors, and female health issues; (2) physical examination results, such as body mass index (BMI), body fat percentage, waist circumference, hip circumference, waist-to-hip ratio, blood pressure, heart rate, pulmonary function, and bone mineral density; (3) blood and urine analyses results from blood tests, serology tests, hepatobiliary function tests, renal function tests, and urinalysis; and (4) data on PAE content of urine

ELIGIBILITY:
inclusion:

1. The target subjects of this study are individuals aged 30 to 70 years old
2. who were tested for PAEs from January 1, 2016 to December 31, 2020.

exclusion:

1who have not been tested for plasticizers

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study included 1337 subjects, with an average age of 48.98 years. Male subjects (51.8%) outnumbered the females. In addition, 75.1% of the subjects were married, 9.4% had drinking habits, 57.4% did not exercise regularly, 15.3% worked in the manufacturing industry, 47.4% were overweight according to BMI, 45.2% had a body fat percentage higher than normal, and 16.8% had bone density below 2.5. Table 1 shows the analysis results.
Sampling Method: Non-Probability Sample
Enrollment: 1136 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Risk assessment analysis of disease and PAEs | 2022
  (1) questionnaire responses, such as basic personal information, individual health behaviors, and female health issues; (2) physical examination results, such as body mass index (BMI), body fat percentage, waist circumference, hip circumference, waist-to-hip ratio, blood pressure, heart rate, pulmonary function, and bone mineral density; (3) blood and urine analyses results from blood tests, serology tests, hepatobiliary function tests, renal function tests, and urinalysis; and (4) data on PAE content of urine.
Artificial intelligence prediction model for diseases and PAEs | 2022
  to apply machine learning to establish the correlations between the environmental hormone PAE and high disease risk and suggest assessment items for nursing intervention.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Cheng Hsin General Hospital, Taipei
  - National Taipei university of nursing and health science, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu HT, Liao CC, Peng CF, Lee TY, Liao PH. Exploring the application of machine learning to identify the correlations between phthalate esters and disease: enhancing nursing assessments. Health Inf Sci Syst. 2024 Dec 29;13(1):10. doi: 10.1007/s13755-024-00324-4. eCollection 2025 Dec. PMID 39736874